CLINICAL TRIAL: NCT01106573
Title: Is There an Association Between the Presence of Diabetes, the Degree of Arterial Stiffness and a New Plasma Marker for Vascular Elasticity, Fibulin-1 in Patients Undergoing Heart- and Vascular Surgery?
Brief Title: Associations Between Diabetes, Arterial Stiffness and Fibulin-1 in Patients Undergoing Heart- and Vascular Surgery?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Odense University hospital
Other Study IDs: KBF2010-01
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Coronary Artery Disease; Arteriosclerosis; Carotid Stenosis; Thrombosis; Aortic Aneurysm, Abdominal
Keywords: Diabetes Mellitus; Arteriosclerosis; Intima media thickness; arterial stiffness; pulsewave velocity; fibulin-1
MeSH Terms: conditions — Coronary Artery Disease; Arteriosclerosis; Carotid Stenosis; Thrombosis; Aortic Aneurysm, Abdominal; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this study we will collect serum, whole blood and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Diabetes Mellitus (DM) is frequently appearing in patients with cardiovascular disease and these patients, as a consequence herby, has a lesser prognosis. DM is often related to increased arterial stiffness and hypertension. The investigators thesis is that DM and pre-diabetes is prevalent in patients undergoing cardiovascular surgery and to some extend is under-diagnosed. At the same time the investigators imagine that DM is closely related to the degree of arterial stiffness, and that these parameters are closely related to a new biochemical marker, fibulin-1.

The investigators aim to describe the prevalence of type 2 DM and dysmetabolism in patients admitted to the hospital to undergo cardiovascular surgery and besides that to investigate if there is a connection between the degree of the dysmetabolism and arterial disease, by studying arterial stiffness and by measuring a new biochemical marker, fibulin-1, which the investigators newly have identified. The results of this project will give us a measure for the quantity of unknown DM in patients undergoing cardiovascular surgery and furthermore tell us more in terms of the connections between a newly identified plasma arterial marker, arterial stiffness and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* undergoing heart- or vascular surgery

Exclusion Criteria:

* Physical or mental disability not enabling participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from patients undergoing planned heart and vascular surgery at our department.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Melholt Rasmussen, Professor, MD, Study Chair — Department of Biochemnistry and Farmacology, Odense University Hospital
Locations (1):
- Department of Biochemnistry and Farmacology, Odense University Hospital, Odense, Denmark